CLINICAL TRIAL: NCT00984555
Title: Assessment of the Vaginal Residence Time of Biomarkers of Semen Exposure
Brief Title: Residence Time of Biomarkers of Semen Exposure
Status: Completed | Type: Observational
Sponsor: CONRAD (Other)
Collaborators: Johns Hopkins University (Other); Eastern Virginia Medical School (Other)
Responsible Party: Jill Schwartz, Medical Director, CONRAD
Other Study IDs: A07-105
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Semen Exposure
Keywords: Biomarkers; Semen Exposure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swabs, semen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A1 (Inoculation with 7 timepoints): Semen exposure via inoculation, Vaginal swabs at 7 time points
- A2 (Inoculation with 4 timepoints): Semen exposure via inoculation, Vaginal swabs at 4 time points
- B1 (intercourse with 7 timepoints): Semen exposure via unprotected intercourse, Vaginal swabs at 7 time points
- B2 (Intercourse with 4 timepoints): Semen exposure via unprotected intercourse, Vaginal swabs at 4 time points

SUMMARY:
The purpose of this study is to examine the vaginal residence time of certain semen biomarkers.

DETAILED DESCRIPTION:
The study will take approximately 2-3 months to complete. First, you will be screened to see if you are eligible for the study. At this visit the male partner will give a medical history and be asked to donate a semen sample for analysis, while the female will give a medical history, receive a physical exam, pelvic exam, pregnancy test, and will be tested for vaginal infection including Gonorrhea/Chlamydia. If you are eligible (as a couple), you will be called and randomized into one of four study groups. You will be allowed to choose whether you want to take certain samples yourself at home, or have them all taken by a nurse at the clinic. At this point you will either be asked to return home to have sexual intercourse, or the male partner will be asked to donate a semen sample, which will then be inserted into the female's vagina. Depending on which group you are in, you will next be asked to return to the clinic either 4 or 7 times over the next 2 weeks for vaginal swabs.

Once you complete the main study, you will be offered the opportunity to participate in a substudy, where you will repeat the same visits, except that if you chose to have all your samples taken in the clinic for the main study, you will take certain samples at home for the substudy. If you chose to take certain samples at home for the main study, you will have all the samples taken at the clinic for the substudy. Also, you will not need to do another screening visit if you start the substudy within 9 weeks of the end of the main study.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual, monogamous couples
* Must not be using birth control other than a tubal ligation
* Must be at least 18 years old, and healthy (if female)
* Must be between 18-55 years old, and healthy (if male)

Exclusion Criteria:

* History of hysterectomy (females)
* History of vasectomy (males)
* Drug or alcohol abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Levels of listed biomarkers in vaginal swabs taken | 6, 24, 48, 72 hours and 7, 11 and 15 days after vaginal inoculation with semen or unprotected intercourse

SECONDARY OUTCOMES:
Percent of all women with a detectable level of each marker at each time point | 6, 24, 48, 72 hours, and 7, 11, and 15 days after vaginal inoculation with semen or unprotected intercourse

CONTACTS AND LOCATIONS:
Overall Officials: Roxanne Jamshidi, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine; David F Archer, MD, Principal Investigator — Eastern Virginia Medical School
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Derived] Thurman A, Jacot T, Melendez J, Kimble T, Snead M, Jamshidi R, Wheeless A, Archer DF, Doncel GF, Mauck C. Assessment of the vaginal residence time of biomarkers of semen exposure. Contraception. 2016 Nov;94(5):512-520. doi: 10.1016/j.contraception.2016.05.012. Epub 2016 May 31. PMID 27259675